CLINICAL TRIAL: NCT00603330
Title: Infusion of Mesenchymal Stem Cells as Treatment for Steroid-Resistant Grade II to IV Acute GVHD or Poor Graft Function: a Multicenter Phase II Study
Brief Title: Mesenchymal Stem Cell Infusion as Treatment for Steroid-Resistant Acute Graft Versus Host Disease (GVHD) or Poor Graft Function
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: KU Leuven (Other); Maastricht University Medical Center (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); University Hospital, Antwerp (Other); University Hospital, Ghent (Other); AZ-VUB (Other); AZ Sint-Jan AV (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital of Mont-Godinne (Other); Jolimont Hospital Haine Saint Paul (Unknown); Queen Fabiola Children's University Hospital (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJB0703P1
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Graft-versus-host Disease; Poor Graft Function; Low Donor T-cell Chimerism
Keywords: Mesenchymal stem cells; Graft-versus-host disease; Poor graft function; Chimerism; Hematopoietic cell transplantation recipients; Low donor T-cell chimerism
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MSC infusion for steroid-refractory grade II-IV acute GVHD. In this arm, 4 x 10E6 MSC/Kg BW of the recipient will be injected during the first hour after thawing.
  Interventions: Biological: Mesenchymal stem cells
- 2 (Experimental): MSC infusion for poor graft function. In this arm, 2 x 10E6 MSC/Kg BW of the recipient will be injected during the first hour after thawing.
  Interventions: Biological: Mesenchymal stem cells
- 3 (Experimental): MSC + DLI for poor donor T-cell chimerism after allogeneic HCT. In this arm, 2 x 10E6 MSC/Kg BW of the recipient will be injected during the first hour after thawing.
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal Stem Cell infusion

SUMMARY:
The present project aims at investigating the role of MSC for the treatment of patients with

Part 1: Steroid-refractory grade II-IV acute GVHD.

Part 2: Poor graft function (PGF)

Part 3: Low or falling donor T-cell chimerism after allogeneic HCT.

This is a multicenter phase II study examining the feasibility and efficacy of this approach.

DETAILED DESCRIPTION:
Part 1: complete recruitment Part 2: complete recruitment Part 3: recruiting

ELIGIBILITY:
Inclusion Criteria:

Patient eligibility criteria

1. Male or female of any age.
2. Previous allogeneic transplantation (related or unrelated donor, any degree of HLA matching) or autologous transplantation (for part 2 only) of HSC at any time before.
3. Any source of HSC (marrow, PBSC, cord blood) and any conditioning regimen.
4. Informed consent given by donor or his/her guardian if of minor age.
5. Additional criteria for each part of the protocol:

Part 1: MSC for steroid-refractory grade II-IV acute GVHD

1. Allogeneic transplantation.
2. Grade II-IV acute GVHD (see appendix A for acute GVHD grading) de novo or following DLI.
3. Acute GVHD refractory to mPDN 2 mg/kg/day or equivalent, defined as

   * progression of GVHD on day 3 after initiation of steroids
   * no improvement of GVHD on day 7 after initiation of steroids
   * absence of complete resolution of acute GVHD on day 14 after initiation of steroids
   * relapse of acute GVHD during or after steroid taper.
4. Ongoing therapy with Ciclosporine or Tacrolimus at therapeutic doses.
5. Patient may have received previously any other form of treatment for acute GVHD, but no new treatment started within 1 month of study entry.

Part 2: MSC for poor graft function (PGF)

1. Allogeneic or autologous transplantation.
2. Cytopenia in 2 or 3 lineages:

   * Hb < 8.0 g/dL and reticulocytes < 1%, with or without transfusion
   * Plt < 20,000/µL without transfusion
   * Neutrophils < 500/µL, without G-CSF administration

   OR severe cytopenia in 1 lineage:
   * RBC transfusion dependent (if autologous transplantation; despite EPO administration if allogeneic transplantation)
   * Plt transfusion dependent
   * Neutrophils < 500/µL despite G-CSF administration
3. Cytopenia duration ≥ 2 weeks beyond day 28 after autologous HCT, or day 42 (day 60 for cord blood transplantation) after allogeneic HCT.
4. Cytopenia is not related to CMV or other infection, myelosuppressive/toxic drugs, renal failure, peripheral cell destruction or other identifiable cause.
5. In case of HLA-identical related donor and full donor chimerism, patient can only be included if a boost of donor CD34+ cells has been unsuccessful or is not feasible.

Part 3: MSC + DLI for poor donor T-cell chimerism

1. Nonmyeloablative allogeneic transplantation.
2. Donor T-cell chimerism < 50% for at least 2 consecutive weeks beyond day 21 after HCT OR

   * 20% decrease in donor T-cell chimerism with the second value < 50%.

MSC donor inclusion criteria

1. Related to the recipient (sibling, parent or child) or unrelated.
2. Male or female.
3. Age > 16 yrs (no age limit if same as HSC donor).
4. No HLA matching required.
5. Fulfills generally accepted criteria for allogeneic HSC donation.
6. Informed consent given by donor or his/her guardian if of minor age.

Exclusion Criteria:

Patient exclusion criteria

1. HIV positive.
2. Active uncontrolled infection at time of scheduled MSC infusion.
3. Relapsing or progressing malignancy.

MSC donor exclusion criteria

1. HIV positive
2. Known allergy to Lidocaine
3. If donor other than HSC donor : any risk factor for transmissible infectious diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Arm 1. Efficacy of MSC infusion as treatment for steroid-resistant grade II - IV acute GVHD. | 30 days
Arm 2. Efficacy of MSC infusion as treatment for poor graft function | 180 days
Arm 3. Efficacy of MSC infusion followed by donor lymphocyte infusion for preventing graft rejection in patients with low or failing donor T-cell chimerism after allogeneic HCT | 180 days

SECONDARY OUTCOMES:
Toxicity of MSC infusion | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Study Chair — CHU-ULg; Frédéric Baron, MD, PhD, Study Chair — CHU-ULg; Johan Maertens, MD, Principal Investigator — KU Leuven; Harry Schouten, MD, Principal Investigator — Maastricht University Medical Center; Pierre Zachée, MD, Principal Investigator — Stuyvenberg Hospital Antwerpen; Zwi Berneman, MD, Principal Investigator — UZA Antwerpen; Lucien Noens, MD, PhD, Principal Investigator — UZ-Gent; Rick Schots, MD, PhD, Principal Investigator — AZ VUB Jette; Dominik Selleslag, MD, Principal Investigator — AZ St. Jan Bugge; Augustin Ferrant, MD, PhD, Principal Investigator — UCL St. Luc Brussels; Chantal Doyen, MD, Principal Investigator — Cliniques Universitaires Mont-Godinne at Yvoir; Nicole Straetmans, MD, Principal Investigator — Hôpital de Jolimont at Haine-St-Paul; Nicole Ferster, MD, Principal Investigator — Hôpital des enfants Reine Fabiola at Brussels
Locations (12):
- Belgium (11):
  - UZA, Edegem, Antwerpen
  - Hôpital des enfants Reine Fabiola, Brussels, Brabant
  - AZ VUB Jette, Brussels, Brabant
  - Cliniques universitaires Saint-Luc- Université Catholique de Louvain, Brussels, Brabant
  - AZ Gasthuisberg Leuven, Leuven, Flamish Brabant
  - UZ Gent, Ghent, Flanders Ost
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - Cliniques Universitaires Mont-Godinne, Yvoir, Namur
  - AZ St Jan, Bruges, West Flanders
  - Hôpital Stuyvenberg, Antwerp
  - CHU Sart Tilman, Liège
- University Hospital Maastricht, Maastricht, Limburg, Netherlands